CLINICAL TRIAL: NCT07330895
Title: Clinical Study of LV009 Injection in the Treatment of Recurrent/Refractory CD19 Positive Blood Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-012-10
Record Dates: First submitted 2025-12-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: CD19+ Relapse/Refractory B-ALL
Keywords: relapse/refractory B-ALL
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- On the Safety, Tolerability, and Efficacy of LV009 Injection in the Treatment of Lymphoma (Experimental): Single dose, single arm trial, exploring the initial 28 day safety and eicacy of the investigational drug.
  Interventions: Drug: Biological: LV009 injection

INTERVENTIONS:
Drug: Biological: LV009 injection — The subjects, who sign the informed consent forms and been screeneinclusion/exclusion criteria, will be assigned into0.3×10^9 TU~2.4×10^9 TU cells.

SUMMARY:
This clinical trial is designed as a single-arm, open-label, single-center investigator-initiated early-phase clinical study, whose primary objective is to evaluate the safety of LV009 Injection in the treatment of subjects with relapsed/refractory CD19-positive hematolymphoid malignancies.

Eligible subjects who have signed the informed consent form will receive an infusion of LV009 Injection. Blood samples will be collected from the subjects before and after the infusion for the evaluation of safety, pharmacokinetics, pharmacodynamics, immunogenicity and other indicators.

In addition to the baseline period, during the treatment phase, efficacy assessments will be conducted at 4 weeks, 2 months, 3 months, 6 months after the infusion of the study drug, and then at a frequency of once every 3 months from the 6th to the 24th month. Tumor assessments will be continued until the occurrence of disease progression (PD), initiation of new anti-tumor therapy, death, intolerable toxicity, decision by the investigator or voluntary withdrawal of the subject, whichever comes first.

DETAILED DESCRIPTION:
All adverse events will be recorded from the start of study drug infusion in subjects until 3 months after drug infusion, disease progression/relapse, initiation of new anti-disease therapy, or study conclusion, whichever comes first. During the period from 3 months after drug administration, disease progression/relapse, or initiation of new anti-disease therapy (whichever occurs first) to the end of the study, only adverse events related to the study product will be collected. Cytokine Release Syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) will be graded according to the Lee Criteria (2019), while all other adverse events (AEs) will be graded based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.

Dose Escalation: A dose escalation study will be conducted according to the designed dose levels. With the exception of the first dose cohort, where only 1 subject will be enrolled from the perspective of benefit-risk assessment and ethics, all other dose cohorts will adopt the traditional "3+3" dose escalation model. Four fixed dose levels of LV009 Injection will be used for escalation, namely: 0.3×10⁹, 0.6×10⁹, 1.2×10⁹, and 2.4×10⁹ Transduction Units (TU).

Dose Escalation Rules: Only 1 subject will be enrolled at the 0.3×10⁹ TU dose level. If a Dose-Limiting Toxicity (DLT) event occurs during the DLT observation period (28 days after cell infusion), the acceleration phase will be terminated and the "3+3" dose escalation study will be initiated. In the "3+3" dose escalation phase, if no DLTs are observed among 3 evaluable subjects, escalation to the next higher dose cohort is permitted. If 1 DLT occurs among 3 evaluable subjects, an additional 3 evaluable subjects need to be enrolled. If ≥1 further DLT occurs (i.e., the total number of subjects with DLT reaches ≥2), the previous dose level will be defined as the Maximum Tolerated Dose (MTD). A total of 10-19 subjects with CD19-positive hematolymphoid malignancies will be enrolled in the study.

Within each dose cohort, the next subject may be administered the study drug only after the previous subject has completed a minimum of 14 days of safety observation. After the last subject in each dose cohort completes the DLT assessment within 28 days following a single administration, enrollment and treatment for the next dose cohort may commence only after the Safety Review Committee (SRC) reviews and approves the move based on the integration of clinical safety data. If 1 DLT occurs among 3 subjects in a dose cohort, 3 additional subjects need to be enrolled in the same dose cohort (resulting in a total of 6 subjects completing DLT assessment in that cohort):

If no DLTs occur in the 3 additional subjects, dose escalation will continue; If 1 DLT occurs in the 3 additional subjects, dose escalation will be terminated; If >1 DLT occurs in the 3 additional subjects, dose escalation will be terminated, and enrollment of 3 additional subjects at one dose level lower will be required for DLT assessment.

If the investigators, through a comprehensive evaluation of the safety, tolerability, and pharmacokinetic data of subjects in a dose cohort, deem it necessary to expand the sample size of that cohort to further observe its safety and pharmacokinetic profile, the cohort may be expanded to a maximum of 6 subjects after reaching a consensus with the sponsor through consultation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of race.
2. Expected survival time exceeds 12 weeks.
3. ECOG score 0-2.
4. Meets the NCCN/CSCO guideline-defined criteria for relapsed/refractory disease and confirmed CD19-positive hematologic malignancy.
5. Liver, kidney, heart, and lung functions meet the following requirements:

   * Creatinine ≤1.5×ULN;
   * Left ventricular ejection fraction ≥45%;
   * Oxygen saturation >91%;
   * Total bilirubin ≤1.5×ULN; ALT and AST ≤2.5×ULN.
6. Absolute lymphocyte count ≥0.5×10⁹/L; platelet count ≥50×10⁹/L; CD3-positive T cells ≥150/uL.
7. Prophylactic anti-allergy medications (e.g., promethazine, diphenhydramine) should be administered 15-30 minutes before investigational drug infusion to prevent cryoprotectant (e.g., DMSO)-related infusion reactions.
8. Subjects must have a body temperature ≤38°C within 24 hours before investigational drug infusion (excluding tumor fever).
9. Within 5 days prior to investigational drug infusion, subjects must not receive therapeutic doses of corticosteroids (>5mg/day prednisone or equivalent) or other immunosuppressive drugs.
10. Before investigational drug infusion, subjects must meet the required washout period per Appendix 3 (Drug/Treatment Discontinuation Schedule). (11) Capable of understanding the trial and having signed informed consent.

Exclusion Criteria:

1. Patients judged by investigators to require long-term use of immunosuppressants during screening.
2. Occurrence of cerebrovascular accident or seizure within 3 months prior to signing informed consent.
3. Presence of other active malignancies besides the studied disease, excluding carcinoma in situ.
4. Peripheral blood hepatitis B virus (HBV) DNA titer exceeding normal reference range.
5. Severe cardiac diseases including but not limited to: unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (NYHA class ≥III), severe arrhythmia.
6. Unstable systemic diseases judged by investigators including but not limited to severe hepatic, renal or metabolic diseases requiring medication.
7. Patients whose acute toxic effects from prior treatment have not yet resolved.
8. Active or uncontrolled infections requiring systemic treatment (excluding mild genitourinary and upper respiratory infections).
9. Female subjects of childbearing potential planning pregnancy within 2 years after investigational drug infusion; or male subjects whose partners plan pregnancy within 2 years after infusion.
10. Prohibited use of investigational drug when following complications exist: clinical evidence of active infection, fluid overload or congestive heart failure, drug-uncontrolled arrhythmia, hypotension requiring vasopressor support.Other situations deemed unsuitable for enrollment/investigational drug infusion by investigators.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 2 years
  Treatment-Emergent Adverse Events (TEAE), Serious Adverse Events (SAE), RCL, and lentiviral integration site status (according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0, NCI CTCAE v5.0)

IPD SHARING:
Plan to Share IPD: No